CLINICAL TRIAL: NCT01274156
Title: The Effect of Low Intensity Shock Wave Therapy on Erectile Dysfunction in Patients Responding to PDE5i's
Brief Title: Double Blind Placebo Controlled Study on the Effect of Extracorporal Shock Wave Therapy on Erectile Dysfunction
Acronym: LI-ESWT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Medispec (Industry)
Responsible Party: Prof Yoram Vardi, Rambam Healthcare Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3060 RMB
Record Dates: First submitted 2010-12-14; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Low Intensity Shock Wave
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- shock wave treatment (Active Comparator)
  Interventions: Device: "MEDISPEC" treatment probe; Device: "MEDISPEC" Low intensity shock waves
- "MEDISPEC" Sham (Sham Comparator): "MEDISPEC" Probe does not deliver energy but creates same noise and sensation of active probe
  Interventions: Device: "MEDISPEC" Sham Probe; Device: Sham

INTERVENTIONS:
Device: "MEDISPEC" treatment probe — 300 shocks in 5 different anatomical locations of the penis.
  Other Names: VASCUSPEC
  Arms: shock wave treatment
Device: "MEDISPEC" Sham Probe — Sham probe applied same as treatment probe without energy
  Other Names: VASCUSPEC
  Arms: "MEDISPEC" Sham
Device: "MEDISPEC" Low intensity shock waves — Treatment parameters will be as follows: Intensity: 0.09 mj/mm2 ,300 shocks per site, on 5 penile anatomical sites. Total number of shock waves: 1500/ session Frequency of 120/min
  Other Names: VASCULOSPEC
  Arms: shock wave treatment
Device: Sham — Probe does not deliver energy but creates same noise and sensation of active probe
  Other Names: Vasculospec
  Arms: "MEDISPEC" Sham

SUMMARY:
This study aims to evaluate the effect of shockwave therapy on erectile dysfunction on patients responding to PDE5i therapy in a sham controlled randomized double blind manner.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of a 12-session low intensity shockwave therapy protocol for patients with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* Rigidity score ≥ 3 under PDE5i therapy
* SHIM ≤21 under PDE5i therapy
* Non- hormonal, neurological or psychological pathology
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Prior prostatectomy surgery
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile function- Erectile Function Domain | At screening and 17 weeks later at last visit
  An increase in score of 5points and above will be considered success.

SECONDARY OUTCOMES:
Rigidity scale | At screening and 17 weeks later at last visit
  A change from 1,2 to a result of 3 or 4 of the rigidity scale points will be considered success
Flow Mediated Dilatation Technique | At screening and 17 weeks later at last visit
  A specialized sphygmomanometer cuff located at the penile base, is inflated to 50 mm Hg for 5min to induce a venous filling. A mercury strain gauge is placed at least 1-2 cm above the penile cuff. Baseline penile blood flow is obtained. Postischemic penile blood flow is then recorded immediately after the deflation, until a return to baseline flow is observed. An increase in blood flow above 30% will be considered success.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel, Israel